CLINICAL TRIAL: NCT05653479
Title: A Randomized, Open-label, Parallel-group, Ethno-bridging Study Comparing the Pharmacokinetics and Safety of a Single Dose of UPB-101 in Healthy Japanese and Non-Japanese Non-East Asian Adults
Brief Title: Safety and Blood Levels After a Single Injection of UPB-101 in Healthy Japanese and Non-Japanese Non-East Asian Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Upstream Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPB-CP-02
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: All treatment groups will enroll and run in parallel. Japanese participants will be enrolled and randomly assigned, on Day 1, to treatment groups 1, 2 or 3. NJNEA participants will be assigned to treatment group 4.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Group 1 (Experimental): Single subcutaneous injection of a low dose of UPB-101 (formerly ASP7266) in 8 Japanese participants
  Interventions: Drug: UPB-101
- Treatment Group 2 (Experimental): Single subcutaneous injection of a medium dose of UPB-101 (formerly ASP7266) in 8 Japanese participants
  Interventions: Drug: UPB-101
- Treatment Group 3 (Experimental): Single subcutaneous injection of a high dose of UPB-101 (formerly ASP7266) in 8 Japanese participants
  Interventions: Drug: UPB-101
- Treatment Group 4 (Experimental): Single subcutaneous injection of a high dose of UPB-101 (formerly ASP7266) in 8 Non-Japanese Non-East Asian participants
  Interventions: Drug: UPB-101

INTERVENTIONS:
Drug: UPB-101 — UPB-101 Subcutaneous injection
  Other Names: Formerly ASP7266

SUMMARY:
The goals of this clinical study are to characterize and compare the safety, tolerability, blood levels of UPB-101 when given to healthy Japanese and non-Japanese non-East Asian (NJNEA) adults. Eligible participants will be assigned to one of the 4 planned dosing treatment groups. Treatment groups 1, 2 and 3 will consist of Japanese adults who will be administered a single subcutaneous (SC) dose of UPB-101 (at 3 different strengths). Treatment group 4 will consist of NJNEA participants who will receive a single SC dose of UPB-101. All treatment groups will enroll and run in parallel.

DETAILED DESCRIPTION:
This is a randomized, open-label, parallel group, ethno-bridging study comparing the pharmacokinetics and safety of a single dose of UPB-101 in healthy Japanese and NJNEA adults. The study will include 4 planned dosing treatment groups. Treatment groups 1, 2 and 3 will consist of Japanese adults who will be administered a single subcutaneous (SC) dose of UPB-101 (at 3 different strengths). Treatment group 4 will consist of NJNEA participants who will receive a single SC dose of UPB-101. All treatment groups will enroll and run in parallel. Japanese participants will be enrolled and randomized on Day 1 into treatment groups 1, 2 or 3 and NJNEA participants will be assigned to treatment group 4.

Eight participants will be enrolled per treatment group, all will receive a single dose of UPB-101. Thus, a total of 32 male and female participants will be enrolled in the study (24 Japanese participants in treatment groups 1-3 and 8 NJNEA participants in treatment group 4).

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female, aged ≥18 to ≤40 years at the date of signing informed consent
2. Body mass index (BMI) between 18 and 25 kg/m2
3. For Japanese (treatment groups 1, 2 and 3), participants must be:

   1. Born in Japan, holding a Japanese passport,
   2. Not living outside Japan for more than 5 years at the date of signing informed consent,
   3. Have all 4 grandparents Japanese

      For NJNEA treatment group 4, participants must be:
   4. Non-Japanese,
   5. Non-East Asian (Chinese, Korean, Mongolian or Taiwanese).
4. Healthy, as defined by:

   1. The absence of clinically significant illness and surgery within 4 weeks prior to dosing.
   2. The absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, haematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
5. Agrees to follow the required contraceptive techniques.
6. Agrees not to donate sperm or ova from the time of the administration of study medication until three months later (120 days)

Main Exclusion Criteria:

1. Current or recurrent disease (or condition), which may put the participant at risk, influence the results of the study, or otherwise affect their ability to participate in the study.
2. Vital signs consistently outside the normal range at Screening or Day -1 and any other abnormal findings or vital signs, ECG, telemetry, physical examination or laboratory evaluation of blood and urine samples that the Investigator judges as likely to interfere with the study or pose an additional risk in participating.
3. Previous exposure or current infection with Hepatitis B, Hepatitis C, tuberculosis (TB), other active recent infection, or history of any untreated or unresolved infection, including parasitic infection.
4. Pregnant or breastfeeding female.
5. Previous exposure to the study drug or known allergy/sensitivity to any of its ingredients.
6. Positive test results for alcohol or drugs of abuse (including cotinine) at Screening or Day -1, or history or clinical evidence of substance and/or alcohol abuse within 2 years before screening.
7. Use of tobacco or other nicotine-containing products in any form within 3 months prior to Day 1.
8. Any recent vaccination, prescription or over-the-counter medication, including herbal remedies or dietary supplements.
9. Recent donation of blood or blood products.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaim Brickman, Study Director — Upstream Bio
Locations (1):
- Richmond Pharmacology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment groups 1, 2, and 3 consisted of Japanese adults who were administered a single SC dose of a low, medium, or high dose of UPB-101, respectively. Treatment group 4 consisted of NJNEA participants who received a single SC dose of a high dose UPB-101.
Groups:
- Low Dose, Japanese: Single subcutaneous injection of a low dose of UPB-101 (formerly ASP7266) in 8 Japanese participants
  UPB-101: UPB-101 Subcutaneous injection
- Medium Dose, Japanese: Single subcutaneous injection of a medium dose of UPB-101 (formerly ASP7266) in 8 Japanese participants
  UPB-101: UPB-101 Subcutaneous injection
- High Dose, Japanese: Single subcutaneous injection of a high dose of UPB-101 (formerly ASP7266) in 8 Japanese participants
  UPB-101: UPB-101 Subcutaneous injection
- High Dose, NJNEA: Single subcutaneous injection of a high dose of UPB-101 (formerly ASP7266) in 8 Non-Japanese Non-East Asian participants
  UPB-101: UPB-101 Subcutaneous injection
Period: Overall Study
Arm/Group | Low Dose, Japanese | Medium Dose, Japanese | High Dose, Japanese | High Dose, NJNEA
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose, Japanese | Medium Dose, Japanese | High Dose, Japanese | High Dose, NJNEA | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (5.66) | 28.6 (5.42) | 31.9 (5.46) | 25.1 (3.68) | 29.2 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 6 | 4 | 15
  Male | 5 | 6 | 2 | 4 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 8 | 8 | 1 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 2
  White | 0 | 0 | 0 | 5 | 5
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 8 | 8 | 8 | 32
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 20.7 (0.81) | 21.2 (1.77) | 20.1 (1.77) | 21.7 (1.73) | 20.9 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of UPB-101
Description: Non-compartmental analysis was used for estimation of PK parameters.
Time Frame: Baseline through Day 85
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Low Dose, Japanese | Medium Dose, Japanese | High Dose, Japanese | High Dose, NJNEA
Number analyzed (Participants) | 8 | 8 | 8 | 8
ug/mL | 11.6 (2.21) | 24.4 (4.77) | 35.1 (12.2) | 34.9 (6.31)

2. Primary Outcome: Time to Maximum Observed Concentration (Tmax) of UPB-101
Description: Non-compartmental analysis was used for estimation of PK parameters.
Time Frame: Baseline through Day 85
Measure: Median (Full Range); unit: days
Arm/Group | Low Dose, Japanese | Medium Dose, Japanese | High Dose, Japanese | High Dose, NJNEA
Number analyzed (Participants) | 8 | 8 | 8 | 8
days | 8.50 [4.0 to 12.0] | 8.00 [5.0 to 12.0] | 8.00 [5.0 to 14.0] | 7.00 [5.0 to 10.0]

3. Primary Outcome: AUC From Time Zero up to the Last Quantifiable Concentration of UPB-101 (AUClast)
Description: Non-compartmental analysis was used for estimation of PK parameters. AUC = Area under the concentration-time curve
Time Frame: Baseline through Day 85
Population: AUClast
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Low Dose, Japanese | Medium Dose, Japanese | High Dose, Japanese | High Dose, NJNEA
Number analyzed (Participants) | 8 | 8 | 8 | 8
day*ug/mL | 407 (88.5) | 755 (84.2) | 1300 (475) | 1200 (235)

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events and Serious Adverse Events
Description: Safety endpoints included AEs, SAEs, physical examinations, clinical laboratory assessments, vital signs, ECGs including telemetry, withdrawal of participants, and early terminations.
Time Frame: Baseline through Day 85
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose, Japanese | Medium Dose, Japanese | High Dose, Japanese | High Dose, NJNEA
Number analyzed (Participants) | 8 | 8 | 8 | 8
Participants | 4 | 4 | 7 | 8

5. Secondary Outcome: Immunogenicity Assessment of UPB-101 When Administered to Japanese and NJNEA Adults
Description: The immunogenicity endpoints included UPB-101 Anti-Drug Antibodies (ADAs). Outcome data is the number of participants with Low titer ADA positive results (range 60-240) observed at Day 85.
Time Frame: Baseline through Day 85
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose, Japanese | Medium Dose, Japanese | High Dose, Japanese | High Dose, NJNEA
Number analyzed (Participants) | 8 | 8 | 8 | 8
Participants | 1 | 3 | 2 | 1

ADVERSE EVENTS:
Time Frame: Baseline through Day 85
Description: Adverse event (AE) data are listed and summarized using descriptive statistics: the number (and %) of participants who had any AEs and the number of AE episodes are summarized by each treatment group
Arm/Group | Low Dose, Japanese | Medium Dose, Japanese | High Dose, Japanese | High Dose, NJNEA
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 4/8 | 7/8 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose, Japanese (N=8) | Medium Dose, Japanese (N=8) | High Dose, Japanese (N=8) | High Dose, NJNEA (N=8)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inner ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (5) | 4 (4)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premenstrual pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT05653479/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT05653479/SAP_001.pdf